CLINICAL TRIAL: NCT03267420
Title: Blood Pressure Measurement: Should Technique Define Targets?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 6486
Record Dates: First submitted 2017-07-20; First posted 2017-08-30 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): A group of 30 randomly assigned study participants that will undergo the BpTRU First, Unattended Omron Second exposure.
  Interventions: Diagnostic Test: BpTRU First, Unattended Omron Second
- Group 2 (Active Comparator): A group of 30 randomly assigned study participants that will undergo the Unattended Omron First, BpTRU Second exposure.
  Interventions: Diagnostic Test: Unattended Omron First, BpTRU Second
- Group 3 (Active Comparator): A group of 30 randomly assigned study participants that will undergo the Partially Attended Omron First, Unattended Omron Second exposure.
  Interventions: Diagnostic Test: Partially Attended Omron First, Unattended Omron Second

INTERVENTIONS:
Diagnostic Test: BpTRU First, Unattended Omron Second — Visit 1: The participants will have the oscillometric device, BpTRU applied to their arm with the higher blood pressure. This will allow assessment with the commonest used Canadian device, which provides an average after 5 unattended readings. This assessment will be followed by the participant wearing a 24 hour ambulatory blood pressure monitor (ABPM) for 24 hours.
  Visit 2: Upon returning the 24 hour ABPM device, the patient will have their blood pressure measured with an unattended Omron second. The Omron HEM 907XL will be applied to the same arm that the BpTRU was applied to in the first visit. There will be 5 minutes of quiet rest (participant alone) and three readings subsequently while the patient is still alone with the average blood pressure measurement being noted.
  Arms: Group 1
Diagnostic Test: Unattended Omron First, BpTRU Second — Visit 1: The participants will have the Omron HEM 907XL will be applied to their arm with the higher blood pressure. There will be 5 minutes of quiet rest (participant alone) and three readings subsequently while the patient is still alone with the average blood pressure measurement being noted.This assessment will be followed by the participant wearing a 24 hour ambulatory blood pressure monitor (ABPM) for 24 hours.
  Visit 2: Upon returning the 24 hour ABPM device, the participants will have the oscillometric device, BpTRU applied to the same arm that the Omron HEM 907 XL was applied to in the first visit. This will allow assessment with the commonest used Canadian device, which provides an average after 5 unattended blood pressure readings.
  Arms: Group 2
Diagnostic Test: Partially Attended Omron First, Unattended Omron Second — Visit 1: The participant will have the Omron HEM 907 XL applied to the arm with the higher blood pressure. There will be five minutes of quiet rest (patient alone) and three reading subsequently, but with the nurse entering the room (i.e., partially attended), with the average being noted. This assessment will be followed by the participant wearing a 24 hour ambulatory blood pressure monitor (ABPM) for 24 hours.
  Visit 2: Upon returning 24 hour ABPM device, the participant will have the Omron HEM 907 XL applied to same arm that was used during the first visit. There will be five minutes of quiet rest (patient alone) and three readings subsequently (patient still alone) with the average blood pressure measurement being noted.
  Arms: Group 3

SUMMARY:
Hypertension is the single most important risk factor for cardiovascular disease and death, yet blood pressure itself is highly influenced by technique and device. Hence, the target blood pressure could vary materially based on BP technique and device used. In the present study, the investigators will compare 4 different methods of measuring blood pressure in the office (casual, resting average of 3 readings with nurse present or absent for resting period, and average of 5 readings) as well as a 24 hour ambulatory measurement. The results of this study will help and enable practicing family physicians and specialists in Canada to target BP for their patients based on algorithm and method of assessment of BP they use in their offices.

DETAILED DESCRIPTION:
Hypertension is the single most important risk factor for cardiovascular disease and death. Over the last several decades many classes of blood pressure lowering drugs have been discovered. These allow physicians to achieve optimal blood pressure and prevent adverse cardiovascular outcomes in most patients. However, the optimal blood pressure level has changed over time, and most recently has been decreased to 120 mm Hg, on the basis of clinical trials. These trials used a specific rigorous method of blood pressure measurement (patient alone in room, enforced period of rest, average of multiple readings) that is currently not the standard of practice in most clinics. Blood pressure itself is highly influenced by technique and device. In particular the length of resting time (if any), and whether it is measured with device requiring medical personnel presence in the room or not. For the same individual, the difference between blood pressure taken with and without rest could be 10 mmHg, and presence vs absence of medical personnel in the room during rest and/or BP assessment could be another 10 mmHg. Hence, the target blood pressure could vary materially based on BP technique and device used. As it is unlikely that all physicians can change their practice overnight and embrace blood pressure device allowing for standard resting time and unattended blood assessment, a comparative pragmatic study of the blood pressure technique and devices endorsed by Hypertension Canada and used in Canada is desirable to avoid either over- or under-treatment of Canadian patients with hypertension.

In the present study, the investigators will compare 4 different methods of measuring blood pressure in the office (casual, resting average of 3 readings with nurse present or absent for resting period, and average of 5 readings) as well as a 24 hour ambulatory measurement in 90 patients. The results of this study will help and enable practicing family physicians and specialists in Canada to target BP for their patients based on algorithm and method of assessment of BP they use in their offices.

ELIGIBILITY:
Inclusion Criteria:

* All patients being followed in the Renal Hypertension Clinic will be eligible for enrollment

Exclusion Criteria:

* Inability to do oscillometric measures (eg., arrhythmia, pain, device reporting error)
* inability to consent the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Casual Blood Pressure versus Omron HEM 907XL unattended | 24 hours: from Visit 1 and Visit 2 (from groups 1, 2 and 3)
  The effect of unattended 5-minute rest preceding unattended systolic blood pressure assessment will be derived from the difference between casual blood pressure (measured in mm Hg) and average resting unattended systolic blood pressure (measured in mm Hg) as measured with the Omron HEM 907 XL

SECONDARY OUTCOMES:
BpTRU versus Omron HEM 907XL with 5 minutes unattended rest | 24 Hours: from Visit 1 and Visit 2 (from groups 1 and 2)
  The difference between average systolic blood pressure measured with BpTRU and Omron HEM907XL (both measured in mm Hg) will allow us to report the effect of the additional five minutes of rest
Omron HEM 907XL unattended versus Omron HEM 907XL partially attended | 24 hours: from Visit 1 and Visit 2 (group 3)
  Difference between systolic blood pressure between the two visits in Group 3 will address an issue of unattended versus partially attended resting systolic blood pressure (both measured in mm Hg)
Omron HEM 907XL unattended versus ABPM device | 24 hours: from Visit 1 and Visit 2 (from groups 1, 2 and 3)
  Difference between the average unattended systolic blood pressure and daytime average blood pressure from the 24 hour ABPM

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Ruzicka, MD, PHD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Hypertension Unit of The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT03267420/Prot_000.pdf